CLINICAL TRIAL: NCT01442701
Title: Stanford's Outcomes Research in Kids (STORK)
Brief Title: Stanford's Outcomes Research in Kids
Acronym: STORK
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Julie Parsonnet, Professor, Stanford University
Other Study IDs: 17756
Record Dates: First submitted 2011-09-01; First posted 2011-09-28 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Bacterial, Viral and Other Infectious Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, skin swabs, stool, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No triclosan / Triclosan: Participants are randomized to receive household and personal cleaning products from one of 2 arms: products that either do not contain triclosan or that may contain triclosan. Participants select products from an arm-specific list of commercially available items.
  Interventions: Other: Removal of triclosan-containing cleaning products from household.

INTERVENTIONS:
Other: Removal of triclosan-containing cleaning products from household. — An intervention is nested within the observational cohort study as a secondary outcome. Commercially available household and personal cleaning products that either do not contain triclosan or that may contain triclosan will be delivered to the household every 4 months for the duration of the study. All cleaning products will be formulated, packaged and labeled by the original manufacturer with no modification for this study. Use of these products will be as per each individual product's label and at the discretion of the participant.

SUMMARY:
The investigators intend to investigate whether the rise in childhood obesity is caused by the loss of recurrent and chronic infections in modern, industrialized society, beginning in utero and extending through early childhood. The investigators will also examine whether the antimicrobial triclosan, present in numerous cleaning and hygiene products, decreases the incidence of infection within a household.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in the study:

1. Able to provide written informed consent.
2. Able to communicate effectively in verbal English or Spanish.
3. Willing to provide blood, saliva, urine and stool specimens from herself, and willing to provide blood, saliva, urine and stool specimens from her infant.
4. Willing to provide consent for review of Primary Provider Medical Records regarding, for the mother, medical history and infectious and other conditions during pregnancy, and for the infant, Apgar scores, height and weight measurements at birth and over time, infectious and other disease diagnoses and treatment, and vaccination records.

Exclusion Criteria:

1. More than one fetus.
2. High risk pregnancy.
3. Intent to move from the Bay Area within three years after enrollment.
4. History of diagnosis and/or treatment, and any current diagnosis or treatment, of type 1 diabetes or of major mental illness.
5. History of diagnosis and/or treatment, and any current diagnosis or treatment, of a thyroid disorder or other endocrine condition.
6. History of diagnosis and/or treatment, and any current diagnosis or treatment that has resulted in severe immunosuppression.
7. A household member who has a compromised immune system
8. Other conditions that in the opinion of the PI would make the subject an unacceptable candidate for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be enrolled from the population of pregnant women attending obstetric clinics for the first antenatal visit. Each woman will be followed throughout her pregnancy and then she and her baby will be followed over the first three years of the baby's life (and more if possible).
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2011-11-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Height-for-weight Z scores | Age 3 years
  We will determine whether an association exists between height-for-weight Z-score (with adjustment for age and sex) and infectious disease load.

SECONDARY OUTCOMES:
Cumulative sick-days | In utero to 3 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ley, PhD, Study Director — Senior Research Scientist
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Background] Ribado JV, Ley C, Haggerty TD, Tkachenko E, Bhatt AS, Parsonnet J. Household triclosan and triclocarban effects on the infant and maternal microbiome. EMBO Mol Med. 2017 Dec;9(12):1732-1741. doi: 10.15252/emmm.201707882. PMID 29030459
- [Background] Ley C, Pischel L, Parsonnet J. Triclosan and triclocarban exposure and thyroid function during pregnancy-A randomized intervention. Reprod Toxicol. 2017 Dec;74:143-149. doi: 10.1016/j.reprotox.2017.09.005. Epub 2017 Sep 20. PMID 28939492
- [Derived] Ley C, Sanchez Mde L, Mathur A, Yang S, Sundaram V, Parsonnet J. Stanford's Outcomes Research in Kids (STORK): a prospective study of healthy pregnant women and their babies in Northern California. BMJ Open. 2016 Apr 13;6(4):e010810. doi: 10.1136/bmjopen-2015-010810. PMID 27075843